CLINICAL TRIAL: NCT04516746
Title: A Phase III Randomized, Double-blind, Placebo-controlled Multicenter Study in Adults, to Determine the Safety, Efficacy, and Immunogenicity of AZD1222, a Non-replicating ChAdOx1 Vector Vaccine, for the Prevention of COVID-19
Brief Title: Phase III Double-blind, Placebo-controlled Study of AZD1222 for the Prevention of COVID-19 in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8110C00001; 2020-005226-28 (EudraCT Number)
Record Dates: First submitted 2020-08-17; First posted 2020-08-18 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind: two or more parties are unaware of the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD1222 (Experimental): Approximately 20,000 participants randomized to the AZD1222 arm
  Interventions: Biological: AZD1222
- Placebo (Placebo Comparator): Approximately 10,000 participants randomized to the saline placebo arm
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AZD1222 — AZD1222 is a recombinant replication-defective chimpanzee adenovirus expressing the SARS-CoV-2-5 surface glycoprotein.
  Arms: AZD1222
Biological: Placebo — Commercially available 0.9% (n/V) saline for injection.
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the safety, efficacy, and immunogenicity of AZD1222 for the prevention of COVID-19.

DETAILED DESCRIPTION:
The COVID-19 pandemic has caused major disruption to healthcare systems with significant socioeconomic impacts. Currently, there are no specific treatments available against COVID-19 and accelerated vaccine development is urgently needed. A safe and effective vaccine for COVID-19 prevention would have significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Increased risk of SARS-CoV-2 infection
* Medically stable

Exclusion Criteria:

* confirmed or suspected immunosuppressive or immunodeficient state
* significant disease, disorder, or finding
* Prior or concomitant vaccine therapy for COVID-19

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32450 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Falsey, MD, Principal Investigator — University of Rochester; Magda Sobieszczyk, MD, Principal Investigator — Columbia University
Locations (74):
- United States (69):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Berkeley, California
  - Research Site, El Centro, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Torrance, California
  - Research Site, Denver, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Coral Gables, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Ankeny, Iowa
  - Research Site, Fairway, Kansas
  - Research Site, Kansas City, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Lake Charles, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Gulfport, Mississippi
  - Research Site, Butte, Montana
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Berlin, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Valhalla, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Yukon, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Sam Houston, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Spring, Texas
  - Research Site, West Jordan, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Fort Belvoir, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, South Charleston, West Virginia
  - Research Site, Madison, Wisconsin
- Chile (2):
  - Research Site, Quillota
  - Research Site, Santiago
- Peru (3):
  - Research Site, Callao
  - Research Site, Lima
  - Research Site, Lima Cercado

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] CDC. (Centers for Disease Control and Prevention). Coronavirus Disease 2019 (COVID-19), Symptoms of Coronavrus. https://www.cdc.gov/coronavirus/2019-ncov/symptomstesting/ symptoms.html. Published 2020. Accessed 01 July 2020.
- [Background] FDA. (Food and Drug Administration). Guidance for Industry. Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. . https://www.fda.gov/media/73679/download. Published 2007. Accessed 20 June 2020.
- [Background] Folegatti PM, Bittaye M, Flaxman A, Lopez FR, Bellamy D, Kupke A, Mair C, Makinson R, Sheridan J, Rohde C, Halwe S, Jeong Y, Park YS, Kim JO, Song M, Boyd A, Tran N, Silman D, Poulton I, Datoo M, Marshall J, Themistocleous Y, Lawrie A, Roberts R, Berrie E, Becker S, Lambe T, Hill A, Ewer K, Gilbert S. Safety and immunogenicity of a candidate Middle East respiratory syndrome coronavirus viral-vectored vaccine: a dose-escalation, open-label, non-randomised, uncontrolled, phase 1 trial. Lancet Infect Dis. 2020 Jul;20(7):816-826. doi: 10.1016/S1473-3099(20)30160-2. Epub 2020 Apr 21. PMID 32325038
- [Background] Li F. Structure, Function, and Evolution of Coronavirus Spike Proteins. Annu Rev Virol. 2016 Sep 29;3(1):237-261. doi: 10.1146/annurev-virology-110615-042301. Epub 2016 Aug 25. PMID 27578435
- [Background] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Background] SPEAC. (Safety Platform for Emergency Vaccines) D2.3 Priority list of adverse events of special interest: COVID-19. Work Package: WP2 Standards and Tools. v1.1. 05 March 2020. https://media.tghn.org/articles/COVID-19_AESIs_SPEAC_V1.1_5Mar2020.pdf. Published 2020. Accessed 14 June 2020.
- [Background] van Doremalen N, Lambe T, Spencer A, Belij-Rammerstorfer S, Purushotham JN, Port JR et al. ChAdOx1 nCoV-19 vaccination prevents SARS-CoV-2 pneumonia in rhesus macaques. bioRxiv. 2020;2020.05.13.093195.
- [Background] Waldrop G, Doherty M, Vitoria M, Ford N. Stable patients and patients with advanced disease: consensus definitions to support sustained scale up of antiretroviral therapy. Trop Med Int Health. 2016 Sep;21(9):1124-30. doi: 10.1111/tmi.12746. Epub 2016 Jul 22. PMID 27371814
- [Background] WHO. (World Health Organization) Coronavirus disease (COVID-19) situation report-175. 13 July 2020. https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200713- covid-19-sitrep-175.pdf?sfvrsn=d6acef25_2. Published 2020. Accessed 13 July 2020.
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Clinical Study Protocol - 1.0 AstraZeneca AZD1222 - D8110C00001 CONFIDENTIAL AND PROPRIETARY 92 of 92
- [Background] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648
- [Derived] Janes H, Fisher LH, Kee JJ, Parameswaran L, Goepfert PA, Falsey AR, Ludwig J, Magaret CA, Gilbert PB, Kublin JG, Rouphael N, Sobieszczyk ME, El Sahly HM, Baden LR, Grinsztejn B, Walsh SR, Gray GE, Kotloff KL, Gay CL, Greninger AL, Tapia MD, Hammershaimb EA, Priddy FH, Green JA, Struyf F, Dunkle L, Neuzil KM, Corey L, Huang Y. Association Between SARS-CoV-2 Viral Load and COVID-19 Vaccination in 4 Phase 3 Trials. J Infect Dis. 2024 Dec 16;230(6):1384-1389. doi: 10.1093/infdis/jiae400. PMID 39225478
- [Derived] Moore M, Zhu Y, Hirsch I, White T, Reiner RC, Barber RM, Pigott D, Collins JK, Santoni S, Sobieszczyk ME, Janes H. Estimating vaccine efficacy during open-label follow-up of COVID-19 vaccine trials based on population-level surveillance data. Epidemics. 2024 Jun;47:100768. doi: 10.1016/j.epidem.2024.100768. Epub 2024 Apr 15. PMID 38643547
- [Derived] Turley CB, Tables L, Fuller T, Sanders LJ, Scott H, Moodley A, Woodward Davis A, Leav B, Miller J, Schoemaker K, Vandebosch A, Sadoff J, Woo W, Cho I, Dunkle LM, Li S, van der Laan L, Gilbert PB, Follmann D, Jaynes H, Kublin JG, Baden LR, Goepfert P, Kotloff K, Gay CL, Falsey AR, El Sahly HM, Sobieszczyk ME, Huang Y, Neuzil KM, Corey L, Grinsztejn B, Gray G, Rouphael N, Luedtke A; COVID-19 Prevention Network CoVPN. Modifiers of COVID-19 vaccine efficacy: Results from four COVID-19 prevention network efficacy trials. Vaccine. 2023 Jul 25;41(33):4899-4906. doi: 10.1016/j.vaccine.2023.06.066. Epub 2023 Jun 23. PMID 37385888
- [Derived] Maaske J, Sproule S, Falsey AR, Sobieszczyk ME, Luetkemeyer AF, Paulsen GC, Riddler SA, Robb ML, Rolle CP, Sha BE, Tong T, Ahani B, Aksyuk AA, Bansal H, Egan T, Jepson B, Padilla M, Patel N, Shoemaker K, Stanley AM, Swanson PA, Wilkins D, Villafana T, Green JA, Kelly EJ. Robust humoral and cellular recall responses to AZD1222 attenuate breakthrough SARS-CoV-2 infection compared to unvaccinated. Front Immunol. 2023 Jan 13;13:1062067. doi: 10.3389/fimmu.2022.1062067. eCollection 2022. PMID 36713413
- [Derived] Aksyuk AA, Bansal H, Wilkins D, Stanley AM, Sproule S, Maaske J, Sanikommui S, Hartman WR, Sobieszczyk ME, Falsey AR, Kelly EJ. AZD1222-induced nasal antibody responses are shaped by prior SARS-CoV-2 infection and correlate with virologic outcomes in breakthrough infection. Cell Rep Med. 2023 Jan 17;4(1):100882. doi: 10.1016/j.xcrm.2022.100882. Epub 2022 Dec 15. PMID 36610390
- [Derived] Sobieszczyk ME, Maaske J, Falsey AR, Sproule S, Robb ML, Frenck RW Jr, Tieu HV, Mayer KH, Corey L, Neuzil KM, Tong T, Brewinski Isaacs M, Janes H, Bansal H, Edwards LM, Green JA, Kelly EJ, Shoemaker K, Takas T, White T, Bhuyan P, Villafana T, Hirsch AI; AstraZeneca AZD1222 Clinical Study Group. Durability of protection and immunogenicity of AZD1222 (ChAdOx1 nCoV-19) COVID-19 vaccine over 6 months. J Clin Invest. 2022 Sep 15;132(18):e160565. doi: 10.1172/JCI160565. PMID 36106642
- [Derived] Falsey AR, Sobieszczyk ME, Hirsch I, Sproule S, Robb ML, Corey L, Neuzil KM, Hahn W, Hunt J, Mulligan MJ, McEvoy C, DeJesus E, Hassman M, Little SJ, Pahud BA, Durbin A, Pickrell P, Daar ES, Bush L, Solis J, Carr QO, Oyedele T, Buchbinder S, Cowden J, Vargas SL, Guerreros Benavides A, Call R, Keefer MC, Kirkpatrick BD, Pullman J, Tong T, Brewinski Isaacs M, Benkeser D, Janes HE, Nason MC, Green JA, Kelly EJ, Maaske J, Mueller N, Shoemaker K, Takas T, Marshall RP, Pangalos MN, Villafana T, Gonzalez-Lopez A; AstraZeneca AZD1222 Clinical Study Group. Phase 3 Safety and Efficacy of AZD1222 (ChAdOx1 nCoV-19) Covid-19 Vaccine. N Engl J Med. 2021 Dec 16;385(25):2348-2360. doi: 10.1056/NEJMoa2105290. Epub 2021 Sep 29. PMID 34587382
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8110C00001&attachmentIdentifier=58e8ea47-f2dc-4d66-bdba-535e1b50a3a3&fileName=D8110C00001_SAP_Redacted.pdf&versionIdentifier=
- See also: D8110C00001-CSP-amendment-6_Redacted.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8110C00001&attachmentIdentifier=90924b91-95c6-4d19-94f1-d5e77e059c8d&fileName=D8110C00001_CSP_Amendment_6_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8110C00001&attachmentIdentifier=a07258a5-fe26-409c-a940-ae25552c538b&fileName=D8110C00001_Clinical_Study_Report_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III randomized study was conducted in adult participants who were healthy or had medically stable chronic diseases and were at increased risk for severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) acquisition and coronavirus disease-2019 (COVID-19) at 88 centers in Chile, Peru and United States of America between 28 August 2020 and 10 February 2023.
Pre-assignment Details: The study had a screening period (14 days), followed by a treatment and follow-up period (up to 760 days). A total of 32450 participants were randomized in a 2:1 ratio to receive AZD1222 or placebo. One participant was enrolled at 2 sites and excluded from all analysis sets. The first participants randomized in each age group in the United States of America participated in a substudy to assess immunogenicity and reactogenicity.
Groups:
- AZD1222: Participants were randomized to receive 2 intramuscular (IM) doses of 5*10^10 viral particles (vp) (nominal, ± 1.5*10^10 vp) AZD1222 on Days 1 and 29.
- Placebo: Participants were randomized to receive 2 IM doses of placebo matching with AZD1222 on Days 1 and 29.
Period: Overall Study
Arm/Group | AZD1222 | Placebo
Started | 21634 | 10816
Participants Who Received First Dose | 21583 | 10797
Participants Who Received Second Dose | 20770 | 9954
Completed | 16099 | 7213
Not Completed | 5535 | 3603
Not completed — Randomized but not Treated | 51 | 19
Not completed — Adverse Event | 0 | 1
Not completed — Death | 62 | 32
Not completed — Lost to Follow-up | 3431 | 1831
Not completed — Withdrawal by Subject | 1946 | 1696
Not completed — Physician Decision | 10 | 8
Not completed — Other | 35 | 16

BASELINE CHARACTERISTICS:
Population: All randomized participants analysis set included all participants who enrolled into the study.
Groups:
- AZD1222: Participants were randomized to receive 2 IM doses of 5*10^10 vp (nominal, ± 1.5*10^10 vp) AZD1222 on Days 1 and 29.
- Total: Total of all reporting groups
Arm/Group | AZD1222 | Placebo | Total
Number analyzed (Participants) | 21634 | 10816 | 32450
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (15.92) | 50.2 (15.86) | 50.2 (15.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9603 | 4797 | 14400
  Male | 12031 | 6019 | 18050
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4787 | 2456 | 7243
  Not Hispanic or Latino | 16506 | 8217 | 24723
  Not reported | 293 | 127 | 420
  Unknown | 48 | 16 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Multiple | 513 | 258 | 771
  White | 17100 | 8534 | 25634
  Black or African American | 1798 | 899 | 2697
  Asian | 947 | 483 | 1430
  American Indian or Alaska Native | 855 | 430 | 1285
  Native Hawaiian or Other Pacific Islander | 60 | 21 | 81
  Not reported | 260 | 138 | 398
  Unknown | 101 | 53 | 154

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Binary Response
Description: A binary response, whereby a participant with negative serostatus at baseline is defined as a COVID-19 case if their first case of SARS-CoV-2 RT-PCR-positive symptomatic illness occurs ≥ 15 days post second dose of study intervention. Otherwise, a participant is not defined as a COVID-19 case. The primary efficacy analysis was performed once approximately 150 events meeting the primary efficacy outcome measure definition had occurred across the AZD1222 and placebo groups.
Time Frame: From 15 days post second dose up to data cut-off date (DCO) of 05 March 2021 or study discontinuation or unblinding or receipt of non-study COVID-19 vaccination, up to a maximum of 17 weeks
Population: The fully vaccinated analysis set (FVS) included all participants in the full analysis set (FAS) who were seronegative at baseline, received 2 doses of study intervention, and who remained on-study 15 days after their second dose without having had a prior SARS-CoV-2 RT-PCR-positive confirmed COVID-19 infection.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 17662 | 8550
Participants | 73 | 130
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; The 95% confidence interval (CI) and p-value were estimated based on Poisson regression with robust variance (including study arm and stratification factor [age group at informed consent] as covariates, and log of the follow up time as an offset); Test type: Superiority; p < 0.001, Poisson regression with robust variance; Vaccine efficacy = 73.98, 95% CI 2-sided [65.34 to 80.47]

2. Primary Outcome: Number of Participants With Adverse Events (AEs) Post Each Dose of Study Intervention
Description: An AE is the development of any untoward medical occurrence in a clinical study participant administered medicinal product and which does not necessarily have a causal relationship with this medicinal product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From Day 1 up to 28 days post second dose of study intervention, approximately 57 days
Population: The safety analysis set included all participants who received at least 1 dose of study intervention from primary analysis data cut which is 1 participant less in placebo group than that from the final data cut.
Measure: Count of Participants; unit: Participants
Groups:
- AZD1222: Participants received 2 IM doses of 5*10^10 vp (nominal, ± 1.5*10^10 vp) AZD1222 on Days 1 and 29.
- Placebo: Participants received 2 IM doses of placebo matching with AZD1222 on Days 1 and 29.
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 21587 | 10792
Participants
  After first dose | 5736 | 1926
  After second dose: number analyzed (Participants) | 20773 | 9947
  After second dose | 5074 | 1797
  After any dose | 8771 | 3201

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAE), Medically Attended Adverse Events (MAAE), and Adverse Event of Special Interest (AESI) Prior to Non-study COVID-19 Vaccination
Description: An SAE is an AE occurring during any study phase that fulfils 1 or more of the following criteria: death; immediately life-threatening; in-participant hospitalization or prolongation of existing hospitalization; persistent or significant disability or incapacity; congenital abnormality or birth defect; an important medical event. AESIs were events of scientific and medical interest specific to the further understanding of the study intervention safety profile and required close monitoring and rapid communication by the investigators to the sponsor. MAAEs are defined as AEs leading to medically-attended visits that were not routine visits for physical examination or vaccination, such as an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Different follow-up time between AZD1222 and Placebo groups (20223 versus 3893 participant years).
Time Frame: From Day 1 up to receipt of non-study COVID-19 vaccination or a maximum of Day 760 for participants without non-study COVID-19 vaccination.
Population: The safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 21587 | 10793
Participants
  SAEs | 621 | 136
  MAAEs | 4750 | 1256
  AESIs | 2516 | 591

4. Primary Outcome: Number of Participants With Local and Systemic Solicited AEs in the Substudy Only
Description: Solicited AEs are local or systemic predefined events for assessment of reactogenicity. Solicited AEs were collected in a e-Diary only for participants in the substudy.
Time Frame: From Day 1 up to 7 days post each dose of study intervention, approximately 14 days
Population: The safety analysis set included all participants who received at least 1 dose of study intervention. Only participants included in the substudy were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 2037 | 1013
Participants
  Solicited local AEs: After first dose: number analyzed (Participants) | 1830 | 920
  Solicited local AEs: After first dose | 1250 | 173
  Solicited local AEs: After second dose: number analyzed (Participants) | 1829 | 908
  Solicited local AEs: After second dose | 977 | 120
  Solicited local AEs: After any dose: number analyzed (Participants) | 1944 | 979
  Solicited local AEs: After any dose | 1440 | 239
  Solicited systemic AEs: After first dose: number analyzed (Participants) | 1842 | 924
  Solicited systemic AEs: After first dose | 1191 | 415
  Solicited systemic AEs: After second dose: number analyzed (Participants) | 1821 | 905
  Solicited systemic AEs: After second dose | 862 | 314
  Solicited systemic AEs: After any dose: number analyzed (Participants) | 1947 | 980
  Solicited systemic AEs: After any dose | 1395 | 519

5. Secondary Outcome: Number of Participants With First Post-intervention Response for SARS-CoV-2 Nucleocapsid Antibodies Post Second Dose of Study Intervention
Description: The incidence of the first post-intervention response (negative at baseline to positive post intervention with study intervention) for SARS-CoV-2 nucleocapsid antibodies occurring ≥ 15 days post second dose of study intervention (key secondary endpoint).
Time Frame: From 15 days post second dose up to DCO of 05 March 2021 or study discontinuation or unblinding or receipt of non-study COVID-19 vaccination, up to a maximum of 17 weeks
Population: The FVS included all participants in the FAS who were seronegative at baseline, received 2 doses of study intervention, and who remained on-study 15 days after their second dose without having had a prior SARS-CoV-2 RT-PCR-positive confirmed COVID-19 infection.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 17662 | 8550
Participants | 156 | 202
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; The 95% CI and p-value were estimated based on Poisson regression with robust variance (including study arm and stratification factor [age group at informed consent] as covariates, and log of the follow up time as an offset); Test type: Superiority; p < 0.001, Poisson regression with robust variance; Vaccine efficacy = 64.32, 95% CI 2-sided [56.05 to 71.03]

6. Secondary Outcome: Number of Participants With First COVID-19 Symptomatic Illness Using Centers for Disease Control and Prevention (CDC) Criteria Post Second Dose of Study Intervention
Description: The incidence of the first case of SARS-CoV-2 RT-PCR-positive symptomatic illness occurring ≥ 15 days post second dose of study intervention using CDC criteria. Participant must present with at least 1 of the following symptoms per CDC criteria: fever, shortness of breath, difficulty breathing, chills, cough, fatigue, muscle aches, body aches, headache, new loss of taste, new loss of smell, sore throat, congestion, runny nose, nausea, vomiting, or diarrhea.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 17662 | 8550
Participants | 95 | 145
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Poisson regression with robust variance; Vaccine efficacy = 69.65, 95% CI 2-sided [60.68 to 76.57]

7. Secondary Outcome: Number of Participants With First COVID-19 Symptomatic Illness Using University of Oxford-Defined Symptom Criteria Post Second Dose of Study Intervention
Description: The incidence of the first case of SARS-CoV-2 RT-PCR-positive symptomatic illness occurring ≥ 15 days post second dose of study intervention using University of Oxford-defined symptom criteria: new onset of fever (> 100 °Fahrenheit [> 37.8 °Celsius]), cough, shortness of breath, or anosmia/ageusia.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 17662 | 8550
Participants | 86 | 136
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Poisson regression with robust variance; Vaccine efficacy = 70.70, 95% CI 2-sided [61.62 to 77.64]

8. Secondary Outcome: Number of Participants With First Symptomatic COVID-19 Regardless of Evidence of Prior SARS-CoV-2 Infection Post Second Dose of Study Intervention
Description: The incidence of the first case of SARS-CoV-2 RT-PCR-positive symptomatic illness occurring ≥ 15 days post second dose of study intervention regardless of evidence of prior SARS-CoV-2 infection (key secondary endpoint).
Time Frame: as for outcome 5
Population: The FVS regardless of prior SARS-COV-2 infection included all participants in the FAS who were seronegative at baseline, received 2 doses of study intervention, and who remained on-study 15 days after their second dose.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 18563 | 9031
Participants | 76 | 135
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Poisson regression with robust variance; Vaccine efficacy = 73.68, 95% CI 2-sided [65.13 to 80.13]

9. Secondary Outcome: Number of Participants With COVID-19 Severe or Critical Symptomatic Illness Post Second Dose of Study Intervention
Description: The incidence of SARS-CoV-2 RT-PCR-positive severe or critical symptomatic illness occurring ≥ 15 days post second dose of study intervention. The severity of COVID-19 was evaluated in participants with symptoms of COVID-19. Following are the findings regarding severe of critical symptomatic COVID-19: clinical signs at rest indicative of severe systemic illness; respiratory failure; evidence of shock; significant acute renal, hepatic, or neurologic dysfunction; admission to an intensive care unit; and death (key secondary endpoint).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 17662 | 8550
Participants | 0 | 8
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; The exact 1-sided 97.5% CI and p-value were estimated based on stratified Poisson regression with exact conditional method (including study arm and stratification factor [age group at informed consent] as strata factor and log of total number of participants for each combination of study arm and strata as an offset); Test type: Superiority; p < 0.001, Poisson regression exact conditional; Vaccine efficacy = 100.00, 97.5% CI 1-sided [lower limit 71.62]

10. Secondary Outcome: Number of Participants With COVID-19 Severe or Critical Symptomatic Illness Post First Dose of Study Intervention
Description: The incidence of SARS-CoV-2 RT-PCR-positive severe or critical symptomatic illness occurring post first dose of study intervention. The severity of COVID-19 was evaluated in participants with symptoms of COVID-19. Following are the findings regarding severe of critical symptomatic COVID-19: clinical signs at rest indicative of severe systemic illness; respiratory failure; evidence of shock; significant acute renal, hepatic, or neurologic dysfunction; admission to an intensive care unit; and death.
Time Frame: as for outcome 5
Population: The FAS included all randomized participants who received at least 1 dose of study intervention, irrespective of their protocol adherence and continued participation in the study. Only participants who are seronegative at baseline were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 20589 | 10300
Participants | 5 | 16
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; The 95% CI were estimated based on Poisson regression with robust variance (including study arm and age group at screening (18-65 years, ≥ 65 years) as covariates and log of the follow-up time as an offset); Test type: Superiority; p < 0.001, Poisson regression with robust variance; Vaccine efficacy = 84.97, 95% CI 2-sided [58.97 to 94.50]

11. Secondary Outcome: Number of Participants With COVID-19-Related Emergency Department Visits Post Second Dose of Study Intervention
Description: The incidence of COVID-19-related emergency department visits occurring ≥ 15 days post second dose of study intervention (key secondary endpoint).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 17662 | 8550
Participants | 1 | 9
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.005, Poisson regression with robust variance; Vaccine efficacy = 94.80, 95% CI 2-sided [58.98 to 99.34]

12. Secondary Outcome: Geometric Mean Titers (GMTs) for SARS-CoV-2 Spike (S) and Receptor Binding Domain (RBD) Antibodies as Measured by Meso Scale Discovery (MSD) Serology Assay
Description: The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titer/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titer, where 'n' is the number of participants with titer information.
Time Frame: Baseline (Day 1) and Days 15, 29, 43, 57, 90, 180, 360, and 730
Population: The immunogenicity analysis population included all participants in the safety analysis set who had no protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response. Only participants included in the substudy were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units per milliliter (AU/mL)
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 2008 | 1002
arbitrary units per milliliter (AU/mL)
  S Antibody Titer: Baseline (Day 1) | 53.18 [50.37 to 56.14] | 54.68 [50.10 to 59.69]
  S Antibody Titer: Day 15: number analyzed (Participants) | 1897 | 949
  S Antibody Titer: Day 15 | 1820.10 [1696.48 to 1952.72] | 53.47 [48.88 to 58.50]
  S Antibody Titer: Day 29: number analyzed (Participants) | 1428 | 708
  S Antibody Titer: Day 29 | 5782.09 [5389.88 to 6202.84] | 53.64 [47.98 to 59.97]
  S Antibody Titer: Day 43: number analyzed (Participants) | 1809 | 899
  S Antibody Titer: Day 43 | 24105.87 [22945.04 to 25325.44] | 58.15 [52.68 to 64.18]
  S Antibody Titer: Day 57: number analyzed (Participants) | 1760 | 829
  S Antibody Titer: Day 57 | 19488.64 [18521.81 to 20505.92] | 58.30 [52.35 to 64.94]
  S Antibody Titer: Day 90: number analyzed (Participants) | 1675 | 643
  S Antibody Titer: Day 90 | 14583.30 [13839.22 to 15367.38] | 87.51 [74.78 to 102.42]
  S Antibody Titer: Day 180: number analyzed (Participants) | 1217 | 147
  S Antibody Titer: Day 180 | 7483.04 [6911.35 to 8102.02] | 266.47 [161.19 to 440.49]
  S Antibody Titer: Day 360: number analyzed (Participants) | 874 | 47
  S Antibody Titer: Day 360 | 6686.81 [5779.74 to 7736.24] | 1268.45 [489.80 to 3284.98]
  S Antibody Titer: Day 730: number analyzed (Participants) | 276 | 22
  S Antibody Titer: Day 730 | 186727.78 [154395.93 to 225830.20] | 19093.94 [5685.04 to 64129.44]
  RBD Antibody Titer: Baseline (Day 1) | 133.6 [129.1 to 138.4] | 138.9 [130.9 to 147.3]
  RBD Antibody Titer: Day 15: number analyzed (Participants) | 1897 | 949
  RBD Antibody Titer: Day 15 | 965.0 [897.0 to 1038.1] | 138.6 [130.5 to 147.1]
  RBD Antibody Titer: Day 29: number analyzed (Participants) | 1427 | 708
  RBD Antibody Titer: Day 29 | 5176.6 [4794.8 to 5588.9] | 143.0 [132.4 to 154.3]
  RBD Antibody Titer: Day 43: number analyzed (Participants) | 1809 | 899
  RBD Antibody Titer: Day 43 | 29351.9 [27875.6 to 30906.4] | 145.7 [136.0 to 156.1]
  RBD Antibody Titer: Day 57: number analyzed (Participants) | 1760 | 829
  RBD Antibody Titer: Day 57 | 23840.6 [22614.3 to 25133.3] | 151.6 [140.3 to 163.8]
  RBD Antibody Titer: Day 90: number analyzed (Participants) | 1675 | 643
  RBD Antibody Titer: Day 90 | 17499.9 [16559.1 to 18494.1] | 192.6 [171.0 to 217.0]
  RBD Antibody Titer: Day 180: number analyzed (Participants) | 1217 | 147
  RBD Antibody Titer: Day 180 | 8333.1 [7647.9 to 9079.7] | 481.6 [314.8 to 736.7]
  RBD Antibody Titer: Day 360: number analyzed (Participants) | 874 | 47
  RBD Antibody Titer: Day 360 | 7499.2 [6417.7 to 8763.1] | 1912.3 [839.0 to 4358.5]
  RBD Antibody Titer: Day 730: number analyzed (Participants) | 276 | 22
  RBD Antibody Titer: Day 730 | 276381.8 [227665.9 to 335521.9] | 19319.4 [5290.3 to 70551.9]

13. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for SARS-CoV-2 S and RBD Antibodies as Measured by MSD Serology Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. GMFR was calculated as anti-logarithm of Σ (log base 2 transformed (post-vaccination titer/ pre-vaccination titer)/n). Where 'n' is the number of participants with titer information.
Time Frame: Days 15, 29, 43, 57, 90, 180, 360, and 730
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 1885 | 943
ratio
  S Antibody Titer: Day 15 | 34.28 [31.87 to 36.86] | 0.97 [0.94 to 1.00]
  S Antibody Titer: Day 29: number analyzed (Participants) | 1420 | 706
  S Antibody Titer: Day 29 | 108.35 [99.95 to 117.45] | 0.92 [0.87 to 0.96]
  S Antibody Titer: Day 43: number analyzed (Participants) | 1797 | 894
  S Antibody Titer: Day 43 | 455.38 [425.71 to 487.12] | 1.08 [1.02 to 1.14]
  S Antibody Titer: Day 57: number analyzed (Participants) | 1746 | 823
  S Antibody Titer: Day 57 | 373.44 [348.12 to 400.60] | 1.10 [1.02 to 1.19]
  S Antibody Titer: Day 90: number analyzed (Participants) | 1664 | 638
  S Antibody Titer: Day 90 | 274.05 [255.01 to 294.50] | 1.61 [1.41 to 1.85]
  S Antibody Titer: Day 180: number analyzed (Participants) | 1207 | 146
  S Antibody Titer: Day 180 | 138.44 [125.37 to 152.88] | 3.33 [2.07 to 5.37]
  S Antibody Titer: Day 360: number analyzed (Participants) | 866 | 46
  S Antibody Titer: Day 360 | 121.12 [102.89 to 142.58] | 17.44 [6.75 to 45.07]
  S Antibody Titer: Day 730: number analyzed (Participants) | 273 | 22
  S Antibody Titer: Day 730 | 3506.74 [2808.52 to 4378.55] | 295.66 [89.07 to 981.35]
  RBD Antibody Titer: Day 15 | 7.24 [6.76 to 7.76] | 1.00 [0.98 to 1.02]
  RBD Antibody Titer: Day 29: number analyzed (Participants) | 1419 | 706
  RBD Antibody Titer: Day 29 | 39.01 [36.10 to 42.17] | 1.01 [0.98 to 1.03]
  RBD Antibody Titer: Day 43: number analyzed (Participants) | 1797 | 894
  RBD Antibody Titer: Day 43 | 219.94 [207.28 to 233.37] | 1.05 [1.01 to 1.09]
  RBD Antibody Titer: Day 57: number analyzed (Participants) | 1746 | 823
  RBD Antibody Titer: Day 57 | 178.61 [167.97 to 189.92] | 1.10 [1.04 to 1.16]
  RBD Antibody Titer: Day 90: number analyzed (Participants) | 1664 | 638
  RBD Antibody Titer: Day 90 | 130.46 [122.53 to 138.89] | 1.41 [1.27 to 1.57]
  RBD Antibody Titer: Day 180: number analyzed (Participants) | 1207 | 146
  RBD Antibody Titer: Day 180 | 61.69 [56.27 to 67.62] | 3.13 [2.11 to 4.65]
  RBD Antibody Titer: Day 360: number analyzed (Participants) | 866 | 46
  RBD Antibody Titer: Day 360 | 53.91 [45.86 to 63.37] | 11.18 [4.91 to 25.45]
  RBD Antibody Titer: Day 730: number analyzed (Participants) | 273 | 22
  RBD Antibody Titer: Day 730 | 2103.65 [1706.88 to 2592.64] | 106.35 [29.93 to 377.87]

14. Secondary Outcome: Percentage of Participants With Seroresponse to the S and RBD Antigens of AZD1222 as Measured by MSD Serology Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. The percentage of participants with a post-intervention seroresponse (≥ 4-fold rise in titers from baseline value to 28 days post each dose) to the S and RBD antigens of AZD1222 as measured by MSD serology assay is reported.
Time Frame: Days 15, 29, 43, 57, 90, 180, 360, and 730
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 1885 | 943
percentage of participants
  S Antibody Titer: Day 15 | 89.8 | 1.1
  S Antibody Titer: Day 29: number analyzed (Participants) | 1420 | 706
  S Antibody Titer: Day 29 | 97.1 | 1.6
  S Antibody Titer: Day 43: number analyzed (Participants) | 1797 | 894
  S Antibody Titer: Day 43 | 99.4 | 2.5
  S Antibody Titer: Day 57: number analyzed (Participants) | 1746 | 823
  S Antibody Titer: Day 57 | 99.3 | 3.2
  S Antibody Titer: Day 90: number analyzed (Participants) | 1664 | 638
  S Antibody Titer: Day 90 | 99.3 | 8.9
  S Antibody Titer: Day 180: number analyzed (Participants) | 1207 | 146
  S Antibody Titer: Day 180 | 98.3 | 23.3
  S Antibody Titer: Day 360: number analyzed (Participants) | 866 | 46
  S Antibody Titer: Day 360 | 96.1 | 54.3
  S Antibody Titer: Day 730: number analyzed (Participants) | 273 | 22
  S Antibody Titer: Day 730 | 100.0 | 90.9
  RBD Antibody Titer: Day 15 | 61.3 | 0.4
  RBD Antibody Titer: Day 29: number analyzed (Participants) | 1419 | 706
  RBD Antibody Titer: Day 29 | 92.2 | 1.0
  RBD Antibody Titer: Day 43: number analyzed (Participants) | 1797 | 894
  RBD Antibody Titer: Day 43 | 98.8 | 2.0
  RBD Antibody Titer: Day 57: number analyzed (Participants) | 1746 | 823
  RBD Antibody Titer: Day 57 | 98.7 | 2.6
  RBD Antibody Titer: Day 90: number analyzed (Participants) | 1664 | 638
  RBD Antibody Titer: Day 90 | 98.6 | 7.7
  RBD Antibody Titer: Day 180: number analyzed (Participants) | 1207 | 146
  RBD Antibody Titer: Day 180 | 96.3 | 22.6
  RBD Antibody Titer: Day 360: number analyzed (Participants) | 866 | 46
  RBD Antibody Titer: Day 360 | 89.8 | 50.0
  RBD Antibody Titer: Day 730: number analyzed (Participants) | 273 | 22
  RBD Antibody Titer: Day 730 | 99.3 | 86.4

15. Secondary Outcome: GMTs for SARS-CoV-2 Neutralizing Antibodies as Measured by Pseudo-neutralization Assay
Description: as for outcome 12
Time Frame: Baseline (Day 1) and Days 15, 29, 43, 57, 90, 180, and 360
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 1943 | 973
AU/mL
  Baseline (Day 1) | 20.6 [20.3 to 20.9] | 21.4 [20.7 to 22.0]
  Day 15: number analyzed (Participants) | 1747 | 920
  Day 15 | 41.7 [39.3 to 44.2] | 21.7 [20.9 to 22.4]
  Day 29: number analyzed (Participants) | 1227 | 682
  Day 29 | 65.9 [60.8 to 71.4] | 23.0 [21.8 to 24.3]
  Day 43: number analyzed (Participants) | 1642 | 876
  Day 43 | 221.3 [208.4 to 235.0] | 22.6 [21.6 to 23.5]
  Day 57: number analyzed (Participants) | 1469 | 777
  Day 57 | 251.8 [235.7 to 269.0] | 23.3 [22.1 to 24.6]
  Day 90: number analyzed (Participants) | 60 | 21
  Day 90 | 206.1 [150.3 to 282.6] | 37.5 [15.0 to 94.1]
  Day 180: number analyzed (Participants) | 283 | 127
  Day 180 | 112.9 [90.4 to 141.0] | 51.3 [37.4 to 70.4]
  Day 360: number analyzed (Participants) | 27 | 14
  Day 360 | 265.7 [94.0 to 751.1] | 46.3 [20.1 to 106.4]

16. Secondary Outcome: GMFR for SARS-CoV-2 Neutralizing Antibodies as Measured by Pseudo-neutralization Assay
Description: as for outcome 13
Time Frame: Days 15, 29, 43, 57, 90, 180, and 360
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 1705 | 896
ratio
  Day 15 | 2.03 [1.92 to 2.15] | 1.01 [0.99 to 1.03]
  Day 29: number analyzed (Participants) | 1200 | 670
  Day 29 | 3.24 [2.99 to 3.50] | 1.07 [1.02 to 1.11]
  Day 43: number analyzed (Participants) | 1597 | 854
  Day 43 | 10.91 [10.27 to 11.58] | 1.05 [1.01 to 1.08]
  Day 57: number analyzed (Participants) | 1432 | 759
  Day 57 | 12.32 [11.54 to 13.16] | 1.08 [1.03 to 1.14]
  Day 90: number analyzed (Participants) | 60 | 20
  Day 90 | 9.95 [7.33 to 13.51] | 1.94 [0.74 to 5.09]
  Day 180: number analyzed (Participants) | 274 | 123
  Day 180 | 5.37 [4.30 to 6.71] | 2.22 [1.65 to 3.00]
  Day 360: number analyzed (Participants) | 26 | 14
  Day 360 | 12.64 [4.31 to 37.11] | 2.31 [1.01 to 5.32]

17. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 Neutralizing Antibodies of AZD1222 as Measured by Pseudo-neutralization Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. The percentage of participants with a post-intervention seroresponse (≥ 4-fold rise in titers from baseline value to 28 days post each dose) to SARS-CoV-2 neutralizing antibodies of AZD1222 as measured by pseudo-neutralization assay is reported.
Time Frame: Days 15, 29, 43, 57, 90, 180, and 360
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 1705 | 896
percentage of participants
  Day 15 | 24.8 | 0.3
  Day 29: number analyzed (Participants) | 1200 | 670
  Day 29 | 41.1 | 1.8
  Day 43: number analyzed (Participants) | 1597 | 854
  Day 43 | 84.4 | 1.9
  Day 57: number analyzed (Participants) | 1432 | 759
  Day 57 | 84.4 | 2.2
  Day 90: number analyzed (Participants) | 60 | 20
  Day 90 | 83.3 | 10.0
  Day 180: number analyzed (Participants) | 274 | 123
  Day 180 | 51.5 | 22.0
  Day 360: number analyzed (Participants) | 26 | 14
  Day 360 | 53.8 | 28.6

18. Secondary Outcome: Number of Participants With COVID-19 Symptomatic Illness Post First Dose of Study Intervention
Description: The incidence of SARS-CoV-2 RT-PCR-positive symptomatic illness occurring post first dose of study intervention.
Time Frame: From Day 1 up to DCO of 05 March 2021 or study discontinuation or unblinding or receipt of non-study COVID-19 vaccination, up to a maximum of approximately 27 weeks
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1222 | Placebo
Number analyzed (Participants) | 20589 | 10300
Participants | 287 | 303
Statistical Analysis 1: Comparison: AZD1222 vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; Vaccine efficacy = 54.47, 95% CI 2-sided [46.48 to 61.26]

ADVERSE EVENTS:
Time Frame: For SAEs: From first dose of study intervention up to 2 years of follow-up post first dose, a maximum of approximately 760 days; For non-serious AEs: From first dose of study intervention up to 28 days post each dose, a maximum of approximately 57 days.
Description: The safety analysis set included all participants who received at least 1 dose of study intervention. Adverse events data reported for double-blind period only. All-cause mortality data reported for overall period (double-blind period and unblinded period).
Arm/Group | AZD1222 | Placebo
All-Cause Mortality (participants affected / at risk) | 62/21587 | 33/10793
Serious Adverse Events (participants affected / at risk) | 1039/21587 | 467/10793
Other Adverse Events (participants affected / at risk) | 11846/21587 | 4234/10793
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1222 (N=21587) | Placebo (N=10793)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Internal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 7 (7) | 4 (4)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Balanitis candida (Infections and infestations) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Device related sepsis (Infections and infestations) | 3 (3) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Monkeypox (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Colon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 6 (7) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Hypobarism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cerebral arteriovenous malformation haemorrhagic (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Osteochondral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Cerebral cavernous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Cerebral palsy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Reactive gastropathy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 2 (2) | 0 (0)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 2 (2) | 0 (0)
Precancerous cells present (Investigations) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 7 (8) | 4 (4)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Renal aplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Thalassaemia minor (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (5)
Limb mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 (16) | 10 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 3 (3)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 7 (7)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Huerthle cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papillary breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 7 (7)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 2 (3)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant splenic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 2 (2)
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (34) | 22 (22)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Retinal melanocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (2)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Alcoholic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Bulbar palsy (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 1 (2) | 2 (3)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 3 (3)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 6 (6) | 3 (3)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Corticobasal degeneration (Nervous system disorders) | 0 (0) | 1 (1)
Delayed myelination (Nervous system disorders) | 1 (2) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 3 (3) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0)
Hemianopia homonymous (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 3 (3) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Internal capsule infarction (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 15 (15) | 7 (8)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 2 (2)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (2) | 0 (0)
Myelomalacia (Nervous system disorders) | 1 (2) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonic epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Neurodegenerative disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post stroke seizure (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 2 (3) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 1 (1)
Syncope (Nervous system disorders) | 8 (8) | 4 (4)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 10 (10) | 8 (8)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 15 (17) | 3 (3)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar II disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 3 (3)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Depression suicidal (Psychiatric disorders) | 2 (2) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 2 (4)
Schizophrenia (Psychiatric disorders) | 1 (1) | 2 (2)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 3 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 5 (5) | 5 (6)
Thyroiditis subacute (Endocrine disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 7 (7) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 13 (13) | 6 (7)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Thyrotoxic crisis (Endocrine disorders) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 6 (6) | 4 (4)
Nephropathy toxic (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal aneurysm (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral caruncle (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (6) | 2 (2)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 3 (3)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 29 (32) | 7 (7)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Endocrine ophthalmopathy (Eye disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 13 (14) | 3 (3)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 4 (4)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery haematoma (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 2 (2) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 3 (4) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic cyst (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 3 (3) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 27 (27) | 7 (7)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 9 (9) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (3) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (2)
Pancreatic failure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatolithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 21 (22) | 13 (13)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 12 (13) | 5 (5)
Small intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 3 (3)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 7 (7) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Drowning (General disorders) | 0 (0) | 1 (1)
Brugada syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 5 (5) | 4 (4)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 4 (5) | 0 (0)
Procedural failure (General disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 9 (11) | 6 (9)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 8 (8) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 9 (9) | 3 (3)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 8 (8) | 3 (3)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 4 (4) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 4 (4) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 29 (31) | 11 (11)
Appendicitis perforated (Infections and infestations) | 4 (4) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 20 (23) | 16 (17)
COVID-19 pneumonia (Infections and infestations) | 29 (34) | 21 (23)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 11 (12) | 7 (8)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Congestive cardiomyopathy (Cardiac disorders) | 1 (2) | 1 (1)
Cholecystitis infective (Infections and infestations) | 2 (2) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 2 (2) | 0 (0)
Colonic abscess (Infections and infestations) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 25 (26) | 5 (7)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 3 (3)
Diverticulitis (Infections and infestations) | 7 (9) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 3 (4) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 3 (4) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Extradural abscess (Infections and infestations) | 3 (3) | 0 (0)
Focal peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 2 (2) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 12 (12) | 10 (10)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 5 (6) | 5 (5)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (2)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (2)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (2)
Myxomatous mitral valve degeneration (Cardiac disorders) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 32 (36) | 8 (9)
Pneumonia bacterial (Infections and infestations) | 5 (5) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Non-obstructive cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (2) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 5 (5) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0)
Renal cyst infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
SARS-CoV-2 sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 11 (11) | 3 (3)
Sepsis syndrome (Infections and infestations) | 1 (2) | 1 (1)
Septic shock (Infections and infestations) | 5 (5) | 2 (2)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Toxic shock syndrome staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (9) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
West Nile viral infection (Infections and infestations) | 1 (2) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Acquired encephalocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1222 (N=21587) | Placebo (N=10793)
Myalgia (Musculoskeletal and connective tissue disorders) | 1622 (1736) | 278 (296)
Headache (Nervous system disorders) | 3511 (4106) | 996 (1125)
Chills (General disorders) | 2208 (2366) | 248 (264)
Fatigue (General disorders) | 2836 (3250) | 853 (942)
Injection site pain (General disorders) | 3624 (4363) | 532 (595)
Pain (General disorders) | 1857 (2023) | 264 (283)
Pyrexia (General disorders) | 1174 (1209) | 73 (78)
COVID-19 (Infections and infestations) | 6207 (6717) | 2715 (2921)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT04516746/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT04516746/SAP_001.pdf